CLINICAL TRIAL: NCT01389037
Title: Promoting Health Literacy of African Americans With High Blood Pressure
Brief Title: Understanding Health Care Information for African Americans With High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00030713; 1P30NR011409 (NIH)
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
Keywords: African American; High blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Literacy-focused Self-help (Experimental)
  Interventions: Behavioral: Health Literacy-focused Self-help
- Delayed intervention control (Placebo Comparator)
  Interventions: Behavioral: Delayed Intervention Control

INTERVENTIONS:
Behavioral: Health Literacy-focused Self-help — Weekly 2-hour sessions over 6 weeks followed by 12 month follow-up with home blood pressure self monitoring with telephone counseling by community health workers.
  Arms: Health Literacy-focused Self-help
Behavioral: Delayed Intervention Control — Given pamphlets on the importance of high blood pressure control and offered weekly workshops. This group will be offered the intervention at the conclusion of data collection.
  Arms: Delayed intervention control

SUMMARY:
This clinical trial focuses on helping African Americans with high blood pressure to manage their disease. The study will target their ability to read and understand health information (also called health literacy). The research method relies on community participation in equal partnership with the researchers to provide interactive workshops and home blood pressure self-monitoring with the assistance of telephone counseling by community health workers.

DETAILED DESCRIPTION:
The purpose of this study is to develop a culturally sensitive intervention focused on health literacy that is designed to reduce high blood pressure (HBP) in a vulnerable African American (AA) population. A community-based participatory research approach delivered by community health workers (CHW) will be used to address the following specific aims: Aim 1. To examine the effect of health literacy on self-care skills, including HBP knowledge, adherence to HBP and substance abuse treatment recommendations, communication skills, health care utilization, and BP outcomes in AAs with HBP. Aim 2. To conduct a pilot randomized, controlled trial with a delayed intervention control group to test the effectiveness of a health literacy-focused self-help HBP intervention program using CHWs in 100 AAs who reside in Baltimore City.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified as African American aged 18 years or older;
2. Systolic BP >140 and/or Diastolic BP >90 mmHg or SBP >135 and/or DBP >85 mmHg for individuals with diabetes mellitus or chronic kidney disease or on HBP medication; and
3. Has a land-based telephone in the home or a cellular phone.

Exclusion Criteria:

1. Participation in another ongoing trial;
2. Acute and/or terminal condition precluding participation, such as terminal cancer;
3. Hospitalization for stroke, myocardial infarction, coronary artery vascularization in the past 3 months;
4. Recipient of an organ transplant or on kidney dialysis; and
5. Psychiatric diagnosis precluding participation, such as schizophrenia or cognitive impairment as measured by Mini-Mental State Exam (score < 24)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Decreased blood pressure | 12 months

SECONDARY OUTCOMES:
Increase adherence to recommended blood pressure management | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Benita Walton-Moss, DNS, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States